CLINICAL TRIAL: NCT06991426
Title: Effects of a New Creatine Formulation (CreaSafe®) on Kidney Function, Skeletal Muscles, and Cardiopulmonary Function in Athletes and Patients With COPD
Brief Title: Effects of CreaSafe® on Kidney, Muscle, and Cardiopulmonary Function in Athletes and COPD Patients
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Rodolfo de Paula Vieira, Prof. Dr., Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2012/15165-2
Record Dates: First submitted 2025-05-06; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Copd; Athletes
Keywords: creatine; supplementation; kidneys; heart; lungs; hematology
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CreaSafe® creatine (Experimental)
  Interventions: Dietary Supplement: CreaSafe® creatine
- Placebo Group Athletes (Placebo Comparator)
  Interventions: Combination Product: Placebo 0.03 g/kg/day
- CreaSafe® creatine COPD (Experimental)
  Interventions: Dietary Supplement: CreaSafe® creatine
- Placebo Group COPD (Placebo Comparator)
  Interventions: Combination Product: Placebo 0.03 g/kg/day

INTERVENTIONS:
Dietary Supplement: CreaSafe® creatine — Will receive CreaSafe® creatine (0.03 g/kg/day) for 90 days, orally administered diluted in water, every morning (between 7:00 and 9:00 a.m.)
  Arms: CreaSafe® creatine; CreaSafe® creatine COPD
Combination Product: Placebo 0.03 g/kg/day — will receive a placebo (microcrystalline cellulose; 0.03 g/kg/day) for 90 days, orally administered diluted in water, every morning (between 7:00 and 9:00 a.m.)
  Arms: Placebo Group Athletes; Placebo Group COPD

SUMMARY:
Creatine supplementation (CS) offers numerous health benefits, with no proven side effects reported to date. CS positively impacts all organs and systems of the body. However, there is an ongoing effort among several creatine-producing companies to develop increasingly pure creatine formulations that generate fewer renal metabolites. Therefore, this study aims to evaluate the effects of a new creatine formulation, CreaSafe®, synthesized by the Chinese company Wenda®, on kidney function in athletes and patients with chronic obstructive pulmonary disease (COPD), as well as its effects on skeletal muscles and cardiopulmonary function. Regarding the athletes (Study 1), the sample will consist of 80 healthy athletes (40 strength-training athletes and 40 middle- and long-distance runners). Among each group of 40 athletes, 20 will receive CreaSafe® creatine (0.03 g/kg/day), while the other 20 will receive a placebo (microcrystalline cellulose; 0.03 g/kg/day), for 90 days, orally administered in water in the morning (between 7:00 a.m. and 9:00 a.m.). For the COPD patients (Study 2), 60 patients with severe and/or very severe COPD will be recruited. Of these, 30 will receive CreaSafe® creatine (0.03 g/kg/day), while the other 30 will receive placebo (microcrystalline cellulose; 0.03 g/kg/day), also administered orally in water for 90 days in the morning (between 7:00 a.m. and 9:00 a.m.). The supplementation period for both studies will last 90 days, with assessments performed at baseline and after 90 days. Kidney function will be evaluated through urinalysis (Urine Type I), the balance of pro- vs. anti-inflammatory cytokines, and levels of urea, creatine kinase (CK), and creatinine. Body composition will be assessed using octopolar and multifrequency bioimpedance, along with circumference measurements of body segments. Muscle strength of different muscle groups will be assessed using the E-lastic dynamometer. Biomarkers of skeletal muscle degradation and recovery will also be measured in plasma, including CK, lactate dehydrogenase (LDH), urea, myoglobin, and the levels of IL-1beta, IL-4, IL-6, IL-10, TNF-alpha, Atrogin-1, MuRF-1, and GDF-8 (myostatin). Whole blood analysis (erythrocytes, leukocytes, and platelets) will be performed using a fully automated blood analyzer (Sysmex XS 800i). Pulmonary function will be assessed through pre- and post-bronchodilator spirometry, as well as maximal inspiratory (PIMax) and expiratory (PEMax) pressures using a manovacuometer. Cardiovascular function will be evaluated using electrocardiography (ECG) and cardiovascular hemodynamics assessed by impedance cardiography (PhysioFlow). GraphPad Prism 5.0 software will be used for statistical analyses and graph generation. Paired Student's t-tests will be used to compare pre- and post-intervention values within each group, and unpaired Student's t-tests will be used to compare deltas between the CreaSafe® and placebo groups. Statistical significance will be considered at p ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* resistance-trained athletes middle- and long-distance runners severe and/or very severe COPD

Exclusion Criteria:

* Non-athletes and individuals without a diagnosis of COPD

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Plasma Inflammatory Cytokine Concentrations | Baseline and after 90 days of supplementation
  Plasma inflammatory cytokines (IL-1β, IL-4, IL-6, IL-10, TNF-α) will be measured using DuoSet® ELISA kits (R&D Systems, USA). Blood samples will be collected at baseline and after 90 days of supplementation. Unit of Measure: pg/mL.
  Mean and standard deviation within each group; pre- and post-intervention comparisons.

SECONDARY OUTCOMES:
Renal Safety Assessed by Serum and Urinary Biomarkers | Baseline and after 90 days of supplementation
  Renal safety will be assessed by measuring serum and urinary biomarkers using Labtest® kits (Brazil). The following biomarkers will be analyzed: serum creatinine (mg/dL), estimated glomerular filtration rate (eGFR; mL/min/1.73 m²), serum urea (mg/dL), and urinary microalbuminuria (mg/g creatinine). Samples will be collected at baseline and after 90 days of supplementation with CreaSafe®.
  Unit of Measure:
  Creatinine: mg/dL eGFR: mL/min/1.73 m² Urea: mg/dL Microalbuminuria: mg/g creatinine Data Aggregation: Mean and standard deviation within each group, with intra- and intergroup comparisons between pre- and post-intervention values.
Urinalysis Parameters | Baseline and after 90 days of supplementation
  Urinalysis will be conducted using reagent strips to assess the following parameters: blood (positive/negative), bilirubin (mg/dL), urobilinogen (mg/dL), ketones (mg/dL), proteins (mg/dL), nitrite (positive/negative), glucose (mg/dL), leukocytes (positive/negative), ascorbic acid (mg/dL), pH, and urine specific gravity (density; g/mL). Assessments will be performed at baseline and after 90 days of supplementation.
  Data Aggregation: Descriptive analysis of the prevalence for qualitative measures; mean and standard deviation for quantitative measures, with comparisons pre- and post-intervention.
Urinary Cytokine Concentrations | Baseline and after 90 days of supplementation
  Urinary cytokines will be measured using DuoSet® ELISA kits (R&D Systems, USA). The following cytokines will be analyzed: IL-1β, IL-1ra, IL-2, IL-6, IL-10, IFN-β, IFN-γ, and TNF-α. Samples will be collected at baseline and after 90 days of supplementation.Unit of Measure: pg/mL.
  Data Aggregation: Mean and standard deviation within each group, with intra- and intergroup comparisons between pre- and post-intervention values.
Lean Body Mass Assessed by Multifrequency Bioelectrical Impedance | Baseline and after 90 days of supplementation
  Lean body mass will be assessed using an octopolar multifrequency bioelectrical impedance analyzer. Measurements will be performed at baseline and after 90 days of supplementation with CreaSafe®. Unit of Measure: kg Data Aggregation: Mean and standard deviation within each group; pre- and post-intervention comparisons.
Muscle Strength Assessed by Dynamometry | Baseline and after 90 days of supplementation
  Muscle strength in major muscle groups (biceps, triceps, chest, calf, waist, hips, thighs) will be assessed using an E-lastic dynamometer (AVS Projetos®). Measurements will be conducted at baseline and after 90 days of supplementation. Unit of Measure: kgf (kilogram-force) Data Aggregation: Mean and standard deviation within each group; pre- and post-intervention comparisons.
Plasma Markers of Muscle Damage and Recovery | Baseline and after 90 days of supplementation
  Plasma concentrations of creatine kinase (CK), lactate dehydrogenase (LDH), urea, and myoglobin will be measured using standard spectrophotometric biochemical assays. Blood samples will be collected at baseline and after 90 days of supplementation.
  Unit of Measure:
  CK, LDH, urea: U/L Myoglobin: ng/mL Data Aggregation: Mean and standard deviation within each group; pre- and post-intervention comparisons.

CONTACTS AND LOCATIONS:
Locations (1):
- Evangelical University of Goiás, Anápolis, Goiás, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kreider RB, Stout JR. Creatine in Health and Disease. Nutrients. 2021 Jan 29;13(2):447. doi: 10.3390/nu13020447. PMID 33572884